CLINICAL TRIAL: NCT02911103
Title: Deep Brain Stimulation Surgery for Treatment of Focal Hand Dystonia
Brief Title: Deep Brain Stimulation Surgery for Focal Hand Dystonia
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 160166; 16-N-0166
Record Dates: First submitted 2016-09-21; First posted 2016-09-22 (Estimated); Last update posted 2026-01-26 (Actual); Status verified 2026-01-21

CONDITIONS: Dystonia; Focal Dystonia; Musician's Dystonia
Keywords: Electrophysiology; Neurosurgery; Dystonia; Deep Brain Stimulation
MeSH Terms: conditions — Dystonia; Dystonic Disorders; Dystonia, Focal, Task-Specific

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Active (Experimental): single arm study
  Interventions: Procedure: DBS surgery; Device: Medtronic Activa Rechargeable System

INTERVENTIONS:
Procedure: DBS surgery — Unilateral thalamic DBS therapy
Device: Medtronic Activa Rechargeable System — Used for diagnostic purposes.

SUMMARY:
Researchers want to test a procedure called deep brain simulation (DBS) to treat focal hand dystonia (FHD). A device called a neurostimulator is placed in the chest. It is attached to wires placed in brain areas that affect movement. Stimulating these areas can help block nerve signals that cause abnormal movements.

Objectives:

To test DBS as treatment for FHD. To learn about brain and nerve cell function in people with dystonia.

Eligibility:

People ages 18 and older with severe FHD who have tried botulinum toxin treatment at least twice

Design:

Participation lasts 5 years.

Participants will be screened with:

Medical history

Physical exam

Videotape of their dystonia

Blood, urine, and heart tests

Brain MRI scan

Chest X-ray

Neuropsychological tests: answering questions, doing simple actions, and taking memory and thinking tests.

Hand movement tests

Participants will have surgery: A frame fixes their head to the operating table. A small hole is made in the skull. Wires are inserted to record brain activity and stimulate the brain while they do simple tasks. The wires are removed and the DBS electrode is inserted into the hole. The neurostimulator is placed under the skin of the chest, with wires running to the electrode in the brain. They will have CT and MRI scans during surgery.

Participants will recover in the hospital for about 1 week.

The neurostimulator will be turned on 1 4 weeks after discharge. Participants will have regular visits until the study ends. Visits include:

Checking symptoms and side effects

MRI

Movement, thinking, and memory tests

If the neurostimulator s battery runs out, participants will have surgery to replace it.

DETAILED DESCRIPTION:
Objectives

To confirm the safety and possible trends toward efficacy of thalamic deep brain stimulation (DBS) targeting the ventralis oralis anterior/ventralis oralis posterior (VOA/VOP) nuclear complex in the treatment of subjects with focal hand dystonia (FHD); and to study the electrophysiologic properties of neurons in the VOA/VOP complex. DBS is FDA approved for Parkinson s disease, Essential tremor, Dystonia (humanitarian exemption), Obsessive- Compulsive disorder (humanitarian exemption) but not for focal hand dystonia.

Study population

Five adults with focal hand dystonia will be studied.

Design

This is a pilot study of 5 subjects with severe intractable FHD whose activities of daily living and quality of life are severely impaired. They will be recruited from our clinic and from referring practices. The subjects will undergo unilateral VOA/VOP DBS implantation, followed by programming to optimal parameters. The subjects will be followed at monthly intervals for 3 months, then every 3 months for 2 years, and then every 6 months until 5 years from the start. The safety of the procedure will be the primary outcome of the study. Trends toward efficacy will be assessed in several secondary outcomes, the most important ones being the change in dystonia severity and a quality of life scores. The electrophysiologic features of the motor ventral thalamic neurons will be recorded intraoperatively.

Outcome measures

Primary

-Number and severity of adverse events in the 5-year follow-up period.

Secondary

* Upper extremity sub-score of the Burke-Fahn-Marsden (BFM) scale and Arm Dystonia Disability Scale (ADDS) at baseline and every follow up visit
* For subjects with FHD type musician s dystonia: Tubiana and Chamagne scale at every follow up visit
* For subjects with FHD type Writer s cramp: Writer s Cramp Impairment Scale
* Improvement on patient reported outcomes evaluated by the SF-12 Health Status Survey at baseline and at every follow up visit
* Neuropsychological evaluation at baseline, 3 and 12 months post DBS surgery
* Dose of botulinum toxin injection required at baseline, 1 and 5 years.

Exploratory

* Intraoperatory electrophysiologic characteristics of the motor ventral thalamic neurons
* Local field potentials and their response to stimulation (in participants with implanted pulse generator capable of sensing capabilities)

ELIGIBILITY:
* INCLUSION CRITERIA:
* FHD diagnosed by a neurologist
* BFM upper extremity subscore of 3 or more (score range 0 to 4) or ADDS difficulty of performing score equal to or more than 3.
* Patients must score 3 or below on the Tubiana and Chamagne scale or inability to perform at the concert level or patients must score a rating of "severe" on at least one item, impacting the patient s employment or essential activities on the Writer s Cramp Impairment scale.
* Symptoms causing significant impairment in quality of life and work or daily activities by patient self-assessment and SF12 scale, as reported by subjects. The subjects should be severely impaired in at least one of the following domains: handwriting, typing or playing an instrument. The impairment needs to have affected employment, manifested by substantive change in, or loss of, employment or career of choice.
* All patients must have failed or achieved inadequate benefit (continuing functional impairment) with at least two trials of botulinum toxin treatments.
* Women of childbearing age will have to agree to use contraception methods for the first 3 post operative months.

EXCLUSION CRITERIA:

* Subjects younger than 22 years old.
* MRI findings that would make participation and surgery unsafe (such as tumor or other space occupying lesion, stroke, hemorrhage or hematoma, edema, hydrocephalus, abscess) and MRI findings that would confound study outcomes (such as iron deposits in the basal ganglia, demyelinating disease, traumatic brain injury, structural or developmental abnormality, moderate or severe white matter hyperintensities).
* Subjects with prior brain surgery
* Pregnant or nursing women as safety of DBS has not been established in this group.
* Presence of a more widespread neurologic syndrome with the dystonia being part of it, and/or dystonia caused by an ongoing etiology, such as tardive dystonia associated with ongoing psychotropic treatment or an inherited neurodegenerative syndrome associated with intractable dystonia
* Intellectual disability as measured by the estimated General Ability Index (GAI) of the Wechsler Adult Intelligence Scale 4th Edition (WAIS-IV), which would render the participant not able to provide informed consent or to comply with the study procedures (estimated GAI less than 70)
* Dementia as evidenced by formal neuropsychological evaluation and Mattis Dementia Rating Scale-2 (DRS-2) score below 128.
* Depressed subjects as determined by the neuropsychology or psychiatry screen, including Beck Depression Inventory (BDI) and psychiatric evaluation. Subjects scoring above 20 on the BDI or exhibiting moderate or severe active depression will be excluded
* Subjects with uncontrolled co-existing medical conditions: uncontrolled systemic hypertension with values above 170/100; active heart disease needing immediate intervention; active respiratory disease needing immediate intervention; uncorrected coagulation abnormalities; any condition that would render the patient unable to safely cooperate with the surgery and study tests as judged by the screening physician
* Presence of a contraindication to undergo a brain MRI

  * Metal in the body which would make having an MRI scan unsafe, such as pacemakers, medication pumps, aneurysm clips, metallic prostheses (including metal pins and rods, heart valves or cochlear implants), shrapnel fragments, permanent eye liner or small metal fragments in the eye that welders and other metal workers may have;
  * Uncomfortable in small closed spaces (have claustrophobia) such that the participant will be uncomfortable in the MRI machine;
  * Unable to lay comfortably flat on their back for up to one hour in the MRI scanner;
* Subjects who require diathermy
* Subjects who require post-op MRIs with full body coil

  -- Subjects with an active systematic infection
* Subjects who are immune-compromised
* Subjects who are on anticoagulation therapy that would preclude their ability to undergo the implant procedure
* Subjects who are allergic or have shown hypersensitivity to any materials of the neurostimulation system which may come in contact with the body
* Subjects that cannot appoint a Durable power of attorney (DPA)

Ages: 22 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2029-02-02 (Estimated); Study Completion 2029-02-02 (Estimated)

PRIMARY OUTCOMES:
To confirm the safety of VOA/VOP thalamic DBS in FHD | 5 years
  Number and severity of adverse events in the 5-year follow-up period.

SECONDARY OUTCOMES:
Neuropsychological Evaluation | 5 years
  To perform a neuropsychological evaluation at baseline, 3 and 12 months post DBS surgery of the VOA/VOP complex in subjects with FHD
To determine if thalamic DBS targeting the VOA/VOP nuclear complex results in clinical improvement of severe intractable FHD | 5 years
  Burke-Fahn-Marsden (BFM) scale and Arm Dystonia Disability Scale (ADDS) at baseline and every follow up visit
To determine if thalamic DBS targeting the VOA/VOP nuclear complex results in improved patient reported outcomes | 5 years
  Neuropsychological evaluation at baseline, 3 and 12 months post DBS surgery
To determine if thalamic DBS targeting the VOA/VOP nuclear complex results in improvement of severe intractable FHD in subjects with musician s dystonia | 5 years
  For subjects with FHD type Musician s Dystonia: Tubiana and Chamagne scale at every follow up visit
To determine if thalamic DBS targeting the VOA/VOP nuclear complex results in improvement of severe intractable FHD in subjects with Writer s cramp | 5 years
  For subjects with FHD type writer s cramp: Writer s Cramp Impairment Scale
To evaluate the botulinum toxin dose required for the treatment of FHD at baseline and 1 and 5 years after DBS therapy of the VOA/VOP complex | 5 years
  Dose of Botulinum Toxin at 1 and 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Debra J Ehrlich, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided
It has not been determined whether sharing IPD will be feasible for this study.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2016-N-0166.html